CLINICAL TRIAL: NCT02450747
Title: Performance of a Multifocal Contact Lens - Presbyopia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5692
Record Dates: First submitted 2015-04-17; First posted 2015-05-21 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-11

CONDITIONS: Presbyopia
Keywords: Visual Acuity
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multifocal Test Contact Lens (Experimental): Subjects will wear the etafilcon A Multifocal test lens in a daily wear modality.
  Interventions: Device: etafilcon A MULTIFOCAL

INTERVENTIONS:
Device: etafilcon A MULTIFOCAL — Subjects will wear the test lens for four weeks.

SUMMARY:
This is a four week study to evaluate the performance of a multifocal contact lens in habitual wearers of silicone hydrogel multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males or females age 40 to 70 and has full legal capacity to volunteer.
2. The subject is a current spherical silicone hydrogel multifocal (SiHy) contact lens wearer (defined as a minimum of 2 days per week for at least 6 hours of Daily Wear contact lenses, for a minimum of one month prior to the study) and willing to wear the study lenses on a daily basis (defined as a minimum of 6 hours of wear per day) for the duration of the study.
3. The subject must own a pair of wearable spectacles to wear when they cannot wear the study lenses.
4. The subject's optimal vertexed spherical equivalent distance correction must be between +3.50 and -5.50 Diopters (D) (inclusive) in both eyes.
5. Subjective refraction cylinder power must be less than or equal to 0.75 D in both eyes.
6. Requires a reading addition of +0.75 D to +2.50 D in each eye.
7. The subject must have distance and near visual acuity best correctable to logMAR 0.1 (20/25) or better at both distance and near with subjective refraction for each eye.
8. The subject must read and sign the Informed Consent form.
9. The subject must appear able and willing to adhere the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
2. Participant in unrelated research clinical trial within 30 days prior to enrollment;
3. Known to have any infectious disease (e.g.hepatitis, tuberculosis) or a contagious immunosuppressive disease.
4. Women who are pregnant or lactating or planning a pregnancy at the time of enrollment;
5. Ocular or systemic allergies or disease which might interfere with contact lens wear;
6. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes.
7. Systemic disease or use of medication which might interfere with contact lens wear;
8. Any corneal distortion;
9. Has any known active* ocular disease and/or infection;
10. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable; and only uses rewetting drops on an occasional basis( greater than 2 times per week).
11. Is a habitual monovision contact lens wearer wearing contact lenses on extended wear basis or for the past 6 months;
12. Diagnosed with Diabetes;
13. Is aphakic; or Has entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
14. Has undergone refractive error surgery;
15. Has amblyopia or strabismus;
16. Has anisometropia >2 D between both eyes;
17. Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study;
18. Any grade 3.0 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Efron classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear;
19. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-four (44) subjects were enrolled in this study. Five (5) subjects did not meet the eligibility and were not dispensed a study article. Of the 39 subjects dispensed study lenses all subjects completed the study without any major protocol deviations.
Groups:
- Multi-focal(Etafilcon A): All subjects worn the Test Contact Lens, Multi-focal (etafilcon A) as daily wear modality over a period of four weeks.
Period: Overall Study
Arm/Group | Multi-focal(Etafilcon A)
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Multi-focal(Etafilcon A): All subjects wore the Test Contact Lens, Multi-focal (etafilcon A) as a daily wear modality over a period of four weeks.
Arm/Group | Multi-focal(Etafilcon A)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Black or African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 33
Region of Enrollment [Number; unit: Participants]
  Canada | 39

OUTCOME MEASURES:

1. Primary Outcome: The Total Grade of Conjunctival Hyperemia
Description: Hyperemia (Redness) was assessed using two different parts of the eye, the Bulbar and the Limbal. Hypemeria was measured using the Efron Scale in 0.5 step units. Grade 0= No Findings, Grade 1= Slight, Grade 2= Mild , Grade 3= Moderate and Grade 4 = severe. Hypermia was assessed in four regions of the eye (Inferior, Nasal, Temporal and Superior). The total grade of Conjunctival Hypermia across all regions and grades is reported. The total grade can range from 0 to 8. Where a higher grade implies worsening conjunctival hypermia
Time Frame: Baseline to 4-Week Follow-up
Population: The analysis population consists of all subjects that completed all study visits without a major protocol deviation. The analysis is conducted on subject eyes.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Subject Eyes
Groups:
- Baseline: Measurements taken at baseline are on all subjects that had already been dispensed the study lens. Only baseline measurements from subject included in the analysis population was reported.
- Multi-focal(Etafilcon A): All subjects wore the study lens, Multi-focal (etafilcon A ) as daily wear modality over a period of four weeks.
Arm/Group | Baseline | Multi-focal(Etafilcon A)
Number analyzed (Participants) | 39 | 39
Number analyzed (Subject Eyes) | 78 | 78
units on a scale
  Bulbar | 4.25 (1.261) | 3.72 (1.232)
  Limbal | 3.51 (1.222) | 3.42 (1.332)

2. Primary Outcome: Upper Lid Margin Staining Score
Description: Upper Lid Margin Staining was assessed using Fluorescein Staining and was measured on the Graded Scale is Grade 0: No Staining is present, Grade 1= 1% to 25% Stains, Grade 2= 26% to 50% Stains, Grade 3= 51% to 75% Stains, Grade 4 76% to 100% Stains. The percentage of eyes with upper lid margin staining for each Grade is reported.
Time Frame: Baseline to 4-Week Follow-up
Population: The analysis population consists of all subjects that completed all study visits without a major protocol deviation. The analysis was conducted on subject eyes.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Subject Eyes
Groups:
- Basline: Measurements taken at baseline are on all subjects that had already been dispensed the study lens. Only baseline measurements from subject included in the analysis population was reported.
- Multi-focal(Etafilcon A): All subjects wore the study Lens, Multi-focal (etafilcon A) as a daily wear modality over a period of four weeks.
Arm/Group | Basline | Multi-focal(Etafilcon A)
Number analyzed (Participants) | 39 | 39
Number analyzed (Subject Eyes) | 78 | 78
percentage of eyes
  Grade 0- No Staining | 46.2 | 26.9
  Grade 1 - 1% to 25% Staining | 28.2 | 44.9
  Grade 2 - 26% to 50% Staining | 23.1 | 24.4
  Grade 3 - 51% to 75% Staining | 2.6 | 3.9
  Grade 4 - 76% to 100% Staining | 0 | 0.0

3. Primary Outcome: Average Corneal Staining Area Grade
Description: Corneal staining Area Grade was assessed in throughout five (5) regions in the eye (Central, Nasal, Temporal, Inferior, Superior). Corneal Staining was Graded using the Efron scale from 0 to 4 in 0.1 unit steps and converted to a percentage of region that was stained. The average percent of region that was stained was calculated and reported.
Time Frame: Baseline to 4- Week Follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Percentage of Staining
Units Other Than Participants: Subject Eyes
Arm/Group | Baseline | Multi-focal(Etafilcon A)
Number analyzed (Participants) | 39 | 39
Number analyzed (Subject Eyes) | 78 | 78
Average Percentage of Staining
  Central | 0.04 (0.025) | 0.05 (0.297)
  Nasal | 0.08 (0.254) | 0.06 (0.224)
  Inferior | 0.039 (0.590) | 0.28 (0.472)
  Temporal | 0.09 (0.287) | 0.03 (0.203)
  Superior | 0.08 (0.320) | 0.06 (0.228)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- Approximately 7 months
Arm/Group | Multi-focal(Etafilcon A)
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days